CLINICAL TRIAL: NCT04920084
Title: A Pilot Plant-Based Dietary Intervention in Overweight and Obese Patients With Monoclonal Gammopathy of Undetermined Significance (MGUS) and Smoldering Multiple Myeloma (SMM) - The Nutrition Prevention (NUTRIVENTION) Study
Brief Title: A Study of a Plant-Based Diet in People With Monoclonal Gammopathy of Undetermined Significance (MGUS) or Smoldering Multiple Myeloma (SMM)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-135
Record Dates: First submitted 2021-06-04; First posted 2021-06-09 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma
Keywords: Plant-Based Diet; Nutrition; 21-135
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: This is a single-arm, single-center pilot.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plant-based meals (Experimental): Patients who will be administered a whole-foods plant-based diet for 12 weeks with nutrition counselling for 24 weeks.Participants will be asked to complete a survey via MSK Engage and a notification will be sent via email notification.
  Interventions: Other: Plant based meals

INTERVENTIONS:
Other: Plant based meals — For 12 weeks, patients will receive two premade meals per day, for lunch and dinner, prepared and shipped weekly by U.S.-based WFPBD company Plantable. The meals will have a low glycemic index and contain vegetables, whole grains, and plant-based fats that have undergone minimal processing. Instructions will be provided for food storage and reheating. Detailed recommendations for snacks and breakfasts meeting the standard of a WFPBD will also be given to supplement their daily calorie needs with access to an online portal from Plantable which contains education materials and access to a coach daily for 24 weeks.

SUMMARY:
This study will test whether a plant-based diet is practical (feasible) for overweight people with monoclonal gammopathy of undetermined significance (MGUS) or smoldering multiple myeloma (SMM). The researchers will decide how practical the diet is by looking at how much weight participants lose and how well they are able to stick to the diet. The researchers will also determine whether the diet is effective in preventing multiple myeloma in participants. In addition, they will look at how safe the plant-based diet is for participants, and see if the diet affects participants' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥25
* Confirmed diagnosis of MGUS or SMM
* M spike (immunoglobulin) ≥0.2 g/dL or abnormal free light chain ratio with increased level of the appropriate involved light chain
* Secretory disease
* Age ≥18 years
* Willingness to comply with all study-related procedures
* ECOG performance status of 0-3
* Interest to learn to cook plant based recipes

Exclusion Criteria:

* Patients that already follow a whole foods plant based or vegan diet (ovo-lactovegetarian diets are not excluded)
* Legume allergy
* Severe allergies, such as anaphylactic shock to peanuts
* Concurrent participation in weight loss/dietary/exercise programs
* Mental impairment leading to inability to cooperate
* Enrollment onto any other therapeutic investigational study
* Concurrent pregnancy
* Patients with a known diagnosis of diabetes mellitus will not be excluded but will need to be followed regularly with an endocrinologist/primary care physician during the trial period.
* Positive HBV, HCV, HIV PCR testing
* Non English speaking
* ≥ Grade 2 electrolyte abnormalities as defined by CTCAEv5.0 (need to be resolved before enrolling on study)
* If in the opinion of the investigator there maybe any concerns regarding the ability of the patient to complete the study safely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2026-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Urvi A Shah, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Plant-based Meals
Started | 23
Completed | 18
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Plant-based Meals
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 62 [40 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Difference of Body Mass Index From Baseline to Week 12
Description: Weight loss is defined as the average decrease in BMI at 12 weeks
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | Plant-based Meals
Number analyzed (Participants) | 20
kg/m^2
  BMI at baseline | 34.30 [30.52 to 38.50]
  BMI at 12 weeks | 32 [26.7 to 36.82]

2. Primary Outcome: Percentage of Whole Food, Plant-based Diet/WFPBD Meals Consumed at Baseline and at 12 Weeks
Description: Intervention defined as ≥70% of participants consuming a whole food, plant-based diet/WFPBD for ≥70% of meals of the 12-week intervention period (determined via a dietary recall and nutritional survey).
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of WFPBD meals consumed
Arm/Group | Plant-based Meals
Number analyzed (Participants) | 20
percentage of WFPBD meals consumed
  Adherence at baseline | 21 [10 to 38]
  Adherence at 12 weeks | 93 [84 to 96]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Plant-based Meals
All-Cause Mortality (participants affected / at risk) | 1/23
Serious Adverse Events (participants affected / at risk) | 14/23
Other Adverse Events (participants affected / at risk) | 15/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plant-based Meals (N=23)
Small intestinal obstruction (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Febrile autoimmune neutropenia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Indigestion/Dysgeusia (Nervous system disorders) | 2
Polyps (Skin and subcutaneous tissue disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1
Herpes simplex reactivation (Infections and infestations) | 1
Thrush (Infections and infestations) | 1
Shingles (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Skin changes (dry, rash, hyperpigmentation) (Skin and subcutaneous tissue disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 1
Nasal congestion/Rhinorrhea/Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Hot flashes (Vascular disorders) | 2
Anxiety (Psychiatric disorders) | 1
Pain (back/extremity/bone) (Musculoskeletal and connective tissue disorders) | 6
Fatigue/weakness/dizziness/fall (General disorders) | 6
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1
Headache (Nervous system disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plant-based Meals (N=23)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 3
Headache (Nervous system disorders) | 2
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Thrush (Infections and infestations) | 1
Shingles (Infections and infestations) | 1
UTI (Infections and infestations) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hot flashes (Vascular disorders) | 1
Polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Nausea (Gastrointestinal disorders) | 1
Herpes simplex reactivation (Infections and infestations) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Indigestion (Gastrointestinal disorders) | 1
Tooth infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT04920084/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT04920084/ICF_001.pdf